CLINICAL TRIAL: NCT06874868
Title: Assessment of Salivary Cortisol As a Biomarker in Patients with Temporomandibular Disorder
Brief Title: Salivary Cortisol As a Biomarker in Patients with Temporomandibular Disorder
Status: Recruiting | Type: Observational
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Bruno Macedo de Sousa, Professor, University of Coimbra
Other Study IDs: FMUCMD2025
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-09

CONDITIONS: Temporomandibular Joint Disorder
Keywords: Temporomandibular disorders; TMD; Cortisol
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Case group: Control group

SUMMARY:
t is recognized that cortisol, a hormone produced by the adrenal glands, is a marker that is elevated in patients with psychological disorders, particularly anxiety. On the other hand, Temporomandibular Disorders (TMD) are a condition with a multifactorial etiology, in which emotional disturbances play a crucial role.

Therefore, the aim of this study is to evaluate whether patients with TMD have higher levels of salivary cortisol compared to the general population.

Initially, an assessment will be conducted using the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) protocol to determine whether the patient suffer of any kind of Temporomandibular Disorder. Based on the results, individuals will be classified into two groups: the study group, consisting of patients with TMD, and the control group, composed of individuals without the disorder.

Those who agree to participate will be required to sign an informed consent form. Subsequently, a saliva sample will be collected for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who attend the dental clinic of the Faculty of Medicine of University of Coimbra

Exclusion Criteria:

* Pregnant women, minors and non-autonomous individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with any form of temporomandibular disorder (TMD) based on the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Salivary cortisol concentration | One day
  The collection should be performed at the time specified by the physician and at least 30 minutes after the ingestion of solid or liquid foods. A collection tube must be obtained from the laboratory, and the following steps should be followed:
  Remove the smaller tube from the collection kit. Open the tube, take out the swab, and place it in the mouth. Gently chew the swab for approximately 1 minute or until swallowing the accumulated saliva becomes unavoidable.
  Return the swab to the smaller tube, ensure it is securely sealed, and then place it inside the larger tube.
  Immediately freeze the sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine of University of Coimbra, Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macedo de Sousa B, Lopez-Valverde N, Cardoso C, Lopez-Valverde A, Rodrigues MJ, Blanco Rueda JA. Evaluation of the salivary biomarker cortisol in patients with temporomandibular disorders. J Oral Facial Pain Headache. 2026 Jan;40(1):81-87. doi: 10.22514/jofph.2026.007. Epub 2026 Jan 12. PMID 41607325